CLINICAL TRIAL: NCT04299880
Title: A Rollover Study to Provide Continued Access to Napabucasin for Patients Enrolled in Boston Biomedical-sponsored Napabucasin Protocols
Brief Title: Rollover Study to Provide Continued Access to Napabucasin for Patients Enrolled in Boston Biomedical-sponsored Protocols
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BBI608-901; 2019-004753-87 (EudraCT Number)
Record Dates: First submitted 2020-03-05; First posted 2020-03-09 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Oncology
Keywords: Neoplasms; Neoplasms by Site; Digestive System Neoplasms; Pancreatic Neoplasms; Adenocarcinoma; Neoplasms, Glandular and Epithelial; Digestive System Diseases
MeSH Terms: conditions — Neoplasms; Neoplasms by Site; Digestive System Neoplasms; Pancreatic Neoplasms; Adenocarcinoma; Neoplasms, Glandular and Epithelial; Digestive System Diseases | interventions — napabucasin; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Gemcitabine; Nivolumab; Paclitaxel; Irinotecan; Leucovorin; Fluorouracil; Bevacizumab

STUDY DESIGN:
Intervention Model Description: Individual patients will continue to be treated with napabucasin (monotherapy or combination) in accordance with the parent study under which they were enrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Napabucasin monotherapy (Other): Patients in this arm will receive napabucasin administered orally, twice daily
  Interventions: Drug: Napabucasin
- Napabucasin in combination with Gemcitabine and Nab-paclitaxel (Other): Patients in this arm will receive napabucasin administered orally, twice daily in combination with weekly nab-paclitaxel and gemcitabine administered intravenously once weekly, on 3 of every 4 weeks.
  Interventions: Drug: Napabucasin; Drug: Nab-paclitaxel; Drug: Gemcitabine
- Napabucasin in combination with Nivolumab (Other): Patients in this arm will receive napabucasin administered orally, twice daily in combination with biweekly nivolumab 3mg/kg administered intravenously over 60 minutes.
  Interventions: Drug: Napabucasin; Drug: Nivolumab
- Napabucasin in combination with paclitaxel (Other): Patients in this arm will receive napabucasin administered orally, twice daily in combination with weekly paclitaxel administered intravenously once weekly, on 3 of every 4 weeks.
  Interventions: Drug: Napabucasin; Drug: Paclitaxel
- Napabucasin in combination with FOLFIRI (Other): Patients in this arm will receive napabucasin administered orally, twice daily in combination with biweekly FOLFIRI. Addition of bevacizumab, per Investigator choice, will be permissible.
  Interventions: Drug: Napabucasin; Drug: Irinotecan; Drug: Leucovorin; Drug: 5Fluorouracil; Drug: Bevacizumab

INTERVENTIONS:
Drug: Napabucasin — Oral
  Other Names: BBI608; BBI-608; BB608
Drug: Nab-paclitaxel — Intravenous
  Other Names: Abraxane
  Arms: Napabucasin in combination with Gemcitabine and Nab-paclitaxel
Drug: Gemcitabine — Intravenous
  Other Names: Gemzar
  Arms: Napabucasin in combination with Gemcitabine and Nab-paclitaxel
Drug: Nivolumab — Intravenous
  Other Names: Opdivo
  Arms: Napabucasin in combination with Nivolumab
Drug: Paclitaxel — Intravenous
  Other Names: Taxol
  Arms: Napabucasin in combination with paclitaxel
Drug: Irinotecan — Intravenous
  Arms: Napabucasin in combination with FOLFIRI
Drug: Leucovorin — Intravenous
  Arms: Napabucasin in combination with FOLFIRI
Drug: 5Fluorouracil — Intravenous
  Arms: Napabucasin in combination with FOLFIRI
Drug: Bevacizumab — Intravenous
  Arms: Napabucasin in combination with FOLFIRI

SUMMARY:
This is an open-label, multi-center, multi-national, non-randomized rollover study designed to allow continued access to napabucasin for patients who have participated in a Boston Biomedical-sponsored study and are being treated with napabucasin (monotherapy or combination) and who are deriving continued clinical benefit in the parent study at the time of closure.

DETAILED DESCRIPTION:
This is an open-label, multi-center, multi-national, non-randomized rollover study designed to allow continued access to napabucasin for patients who have participated in a Boston Biomedical-sponsored study and are being treated with napabucasin (monotherapy or combination) and who are deriving continued clinical benefit in the parent study at the time of closure. Individual patients will continue to be treated with napabucasin (monotherapy or combination) in accordance with the parent study under which they were enrolled. If the dose was reduced in the parent protocol, the dose of the last visit of the parent study will be used. Patients will be monitored to determine long term safety and tolerability of napabucasin.

ELIGIBILITY:
Inclusion Criteria

1. The patient is currently participating in a BBI-sponsored parent study of napabucasin and must be receiving napabucasin as monotherapy or as part of a combination treatment.
2. Written, signed consent for trial participation must be obtained from the patient appropriately in accordance with applicable International Conference on Harmonisation (ICH) guidelines and local and regulatory requirements prior to the performance of any study specific procedure.
3. Must be ≥18 years of age.
4. Currently has no evidence of progressive disease, as determined by the investigator, during treatment with napabucasin (either as monotherapy or as part of a combination treatment regimen) or are deriving clinical benefit despite disease progression according to Investigator's clinical judgement.
5. Continued ability to swallow and retain orally administered study drug(s) and does not have any clinically significant GI abnormalities that may alter absorption such as malabsorption syndrome.
6. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test at screening.
7. Non-fertile or agree to use an adequate method of contraception while on study and for 6 months following the last dose and not currently nursing; males agree to use an adequate method of contraception while on study and for 3 months following the last dose (Appendix 3).
8. Patients must be accessible for treatment and follow-up. Patients registered on this trial must receive protocol treatment and be followed at their current (parent study) participating center.
9. Patient agrees not to participate in other interventional clinical studies during their participation in this trial. Patients participating in surveys or observational studies are eligible to participate in this study.

Exclusion Criteria

1. Permanent discontinuation of napabucasin in the parent study.
2. Napabucasin dose interruption for >4 weeks between the last dose on the parent study and first dose on the rollover study.
3. Women who are pregnant or breastfeeding. Women should not breastfeed while taking study treatment and for 4 weeks after the last dose of napabucasin. Women undergoing combination backbone therapy should not breast feed while on combination backbone therapy and for the period of time following discontinuation of combination backbone therapy as specified in the parent protocol.
4. Hypersensitivity to napabucasin or one of the excipients.
5. Any active disease condition which would render the protocol treatment dangerous or impair the ability of the patient to receive protocol therapy.
6. Any condition (e.g. psychological, geographical, etc.) that does not permit compliance with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | From first dose until 30 days following last dose of napabucasin
  Adverse Events, including clinically significant laboratory abnormalities, as characterized by type, frequency, severity (as graded by NCI CTCAE version 4.0), seriousness, and relationship to study therapy.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - OHSU Knight Cancer Institute, Portland, Oregon
- Centre Antoine Lacassagne, Nice, France
- Japan (2):
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Kyorin University Hospital, Tokyo
- Taipei Veterans General Hospital, Taipei, Taiwan